CLINICAL TRIAL: NCT00754468
Title: A STUDY OF CRYOSPRAY ABLATIONTM USING SURGICAL RESECTION SPECIMENS TO DETERMINE TREATMENT EFFECT, DEPTH OF INJURY, AND SIDE EFFECTS IN THE ESOPHAGUS (CSA Depth 3)
Brief Title: Study of CryoSpray Ablation(TM)to Determine Treatment Effect, Depth of Injury, and Side Effects in the Esophagus.
Acronym: ESODOI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSA Medical, Inc. (Industry)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-00017
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Barrett's Esophagus; Esophageal Cancer
Keywords: Barrett's Esophagus; Esophageal Cancer; Esophageal Dysplasia; Low Grade Dysplasia; High Grade Dysplasia
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Cryo Spray Ablation (Experimental): cryo spray ablation applied to healthy tissue 4 cycles x 10 seconds
  Interventions: Device: Cryo Spray Ablation
- Group 2: Cryo Spray Ablation (Experimental): cryo spray ablation applied to healthy tissue 2 cycles x20 seconds
  Interventions: Device: Cryo Spray Ablation

INTERVENTIONS:
Device: Cryo Spray Ablation — Cryo Spray Ablation 4 cycles x 10 seconds treatment
  Arms: Group 1: Cryo Spray Ablation
Device: Cryo Spray Ablation — Cryo Spray Ablation 2 cycles x 20 seconds
  Arms: Group 2: Cryo Spray Ablation

SUMMARY:
The purpose of this study is to evaluate the treatment effect, depth of injury, and side effects using technology involving the spray of liquid nitrogen through a catheter (CryoSpray AblationTM, "CSA" or "cryospray therapy") onto healthy tissue via esophagogastroduodenoscopy (EGD) using surgical resection specimens from subjects undergoing esophagectomy.

DETAILED DESCRIPTION:
The proposed study is a single center study consisting of no more than 10 subjects who are undergoing scheduled esophagectomy for reasons unrelated to the study. Subjects will be divided into 2 Groups in a sequential fashion based on the time of enrollment (Subject 1 in Group1, Subject 2 in Group 2, Subject 3 in Group1, Subject 4 in Group 2, etc). Potential study subjects will be referred from clinical practice. After entry into the study with written informed consent, subjects will be scheduled for the EGD with cryospray ablation treatment 7 days prior to the expected esophagectomy date.

All subjects will receive narcotic analgesics to control symptoms.

Endpoints related to pathology will be assessed by two independent reviewers, one from the Institution's Department of Pathology, and one from an independent Pathology lab chosen by the sponsor. The reviewers will evaluate the pathology slides to assess maximal extent of depth of injury, side effects, and pathological changes associated with CSA. All reviewers will be blinded to the treatment conditions of the specimens.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age
* Esophagectomy planned based on clinical situation not related to this study.
* Deemed operable based on institutional criteria.

Exclusion Criteria:

* Pregnant
* Esophageal stricture preventing passage of endoscope or catheter.
* Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines.
* Refusal or inability to give consent.
* Concurrent chemotherapy.
* Prior or concurrent endoscopic ablation therapy within 4 cm from the CSA treatment area including, but not limited to, cryospray therapy, laser treatment, photodynamic therapy, multi-polar electro coagulation, endoscopic mucosal resection, radiofrequency ablation, or argon plasma coagulation.
* Prior radiation therapy which involved the esophagus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afonso Ribeiro, M.D., Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida, United States

REFERENCES:
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Eisen GM, Sandler RS, Murray S, Gottfried M. The relationship between gastroesophageal reflux disease and its complications with Barrett's esophagus. Am J Gastroenterol. 1997 Jan;92(1):27-31. PMID 8995932
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Cash BD, Johnston LR, Johnston MH. Cryospray ablation (CSA) in the palliative treatment of squamous cell carcinoma of the esophagus. World J Surg Oncol. 2007 Mar 16;5:34. doi: 10.1186/1477-7819-5-34. PMID 17367523
- [Background] Pinsonneault C, Fortier J, Donati F. Tracheal resection and reconstruction. Can J Anaesth. 1999 May;46(5 Pt 1):439-55. doi: 10.1007/BF03012943. PMID 10349923
- [Background] Dumot JA. Cryotherapy Ablation for Esophageal HGD or IMCA in High Risk, Non-Surgical Patients. DDW2007 Abstract submission. Cleveland Clinic Foundation (pending publication)
- [Background] Greenwald BD. CryoSpray Ablation of Early Esophageal Cancer. DDW 2007 Abstract submission. University of Maryland Medical Center. (pending publication)
- [Background] Johnston M, Horwhat J, Dubois A, Schoenfeld P. Endoscopic cryotherapy in the swine esophagus: A follow-up study (Abstract). Gastrointestinal Endoscopy 49:AB126, 1999.
- [Background] Johnston MH, Horwhat JD, Haluska, Moses FM. Depth of injury following endoscopic spray cryotherapy: EUS assisted evaluation of mucosal ablation and subsequent healing in the swine model (Abstract). Gastrointestinal Endoscopy 51: AB98, 3462, 2000.
- [Background] Johnston MH. Endoscopic cryotherapy: A new ice age in gastroenterology? Medscape Gastroenterology 2: 187, 2000.
- [Background] Eastone JA, Horwhat D, Haluska O, Mathews J, Johnston M. Cryoablation of swine esophageal mucosa: A direct comparison to argon plasma coagulation (APC) and multipolar electrocoagulation (MPEC) [Abstract] Gastrointestinal Endoscopy 53: A3448, 2001.
- [Background] Johnston MH, Eastone JA, Horwhat JD. Reversal of Barrett's esophagus with cryotherapy [Abstract]. American Journal of Gastroenterology 98(9 Suppl): A30, S11, 2003.
- [Background] Johnston MH, Cash BD, Horwhat JD, Johnston LR, Dykes CA, Mays HS. Cryoablation of Barrett's Esophagus (BE) [Abstract]. Gastroenterology 130 (4, Suppl.2): A640, 2006.
- [Background] Johnston MH, Cash BD, Dykes CA, Mays HS, Johnston LR. Cryoablation of dysplasia in Barrett's Esophagus (BE) and early stage esophageal cancer [Abstract]. Gastrointestinal Endoscopy 63 (5): April, 2006.
- [Background] Ribeiro A, Bejarano P, Livingstone A, Sparling L, Franceschi D, Ardalan B. Depth of injury caused by liquid nitrogen cryospray: study of human patients undergoing planned esophagectomy. Dig Dis Sci. 2014 Jun;59(6):1296-301. doi: 10.1007/s10620-013-2991-4. Epub 2014 Jan 7. PMID 24395381

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Subjects in Group 1 will receive a cryospray applied to healthy tissue for 10 seconds, as measured by the device integrated timer beginning at the point when a sustained cryofrost appears. The cryospray will be repeated four (4) times in sequential fashion for a total of 40 seconds of cryospray therapy.
  CryoSpray Ablation(TM): CSA Medical, Inc. (formerly CryMed Technologies, Inc.) received FDA market clearance for the CSA System (CryoSpray AblationTM System, formally Cryo Ablator System) on April 21, 2006. It is a Class II device "intended to be used as a cryosurgical tool for the destruction of unwanted tissue in the field of general surgery, specifically for endoscopic applications." (K070893) As defined by the FDA, the CSA System is a cryosurgical unit with a liquid nitrogen cooled cryocatheter and accessories used to destroy tissue during surgical procedures by applying extreme cold.
- Group 2: Subjects in Group 2 will receive a cryospray applied to healthy tissue for 20 seconds, as measured by the device integrated timer beginning at the point when a sustained cryofrost appears. The cryospray will be repeated two (2) times in sequential fashion for a total of 40 seconds of cryospray therapy.
  CryoSpray Ablation(TM): CSA Medical, Inc. (formerly CryMed Technologies, Inc.) received FDA market clearance for the CSA System (CryoSpray AblationTM System, formally Cryo Ablator System) on April 21, 2006. It is a Class II device "intended to be used as a cryosurgical tool for the destruction of unwanted tissue in the field of general surgery, specifically for endoscopic applications." (K070893) As defined by the FDA, the CSA System is a cryosurgical unit with a liquid nitrogen cooled cryocatheter and accessories used to destroy tissue during surgical procedures by applying extreme cold.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 48 [22 to 63] | 64 [61 to 66] | 55 [22 to 66]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Depth of Injury
Description: histopathological findings analyzed to determine max depth of injury (mm)
Time Frame: End of Study
Measure: Mean (80% Confidence Interval); unit: millimeters
Units Other Than Participants: tissue samples
Arm/Group | Group 1: Cryo Spray Ablation | Group 2: Cryo Spray Ablation
Number analyzed (Participants) | 4 | 3
Number analyzed (tissue samples) | 4 | 3
millimeters | 4.0 [1.7 to 6.3] | 5.2 [2.5 to 8.3]

2. Secondary Outcome: Side Effects of Subjects Receiving Cryospray Therapy.
Time Frame: End of Study
Measure: Number; unit: side effects
Arm/Group | Group 1: Cryo Spray Ablation | Group 2: Cryo Spray Ablation
Number analyzed (Participants) | 4 | 3
side effects | 2 | 1

ADVERSE EVENTS:
Time Frame: 72 hours post cryotherapy intervention
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 2/4 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=4) | Group 2 (N=3)
odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0) — painful swallowing
pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — mild pain noted after the procedure

LIMITATIONS AND CAVEATS:
single center, small number of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No